CLINICAL TRIAL: NCT00964197
Title: FemmeJock: A Pilot Study to Assess Patient Satisfaction and Improvement of Pelvic Floor Symptoms Using a Pelvic Floor Support Girdle in Women With Uterovaginal Prolapse.
Brief Title: The Purpose of This Study is to Look at Pelvic Support Problems, Also Commonly Known as Pelvic Organ Prolapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FemmeJock
Record Dates: First submitted 2009-07-17; First posted 2009-08-24 (Estimated); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Pelvic Organ Prolapse
Keywords: FemmeJock; Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FemmeJock (Experimental): The participant will be fitted with the girdle. The participant will use the girdle for the next 3 months. The girdle is only to be worn during the daytime during times of physical activity. The length of time you choose to wear it during the day is the patients choice. In two weeks the participant will be asked to fill out a 5 question survey in a follow up visit. The participant will be asked to return 3 months after wearing the FemmeJock girdle and to fill out a 5 question survey, as well as to complete a 20 question survey.
  Interventions: Device: FemmeJock

INTERVENTIONS:
Device: FemmeJock — The participant will be fitted with the girdle. The participant will use the girdle for the next 3 months. The girdle is only to be worn during the daytime during times of physical activity. The length of time you choose to wear it during the day is the patients choice. In two weeks the participant will be asked to fill out a 5 question survey in a follow up visit. The participant will be asked to return 3 months after wearing the FemmeJock girdle and to fill out a 5 question survey, as well as to complete a 20 question survey.

SUMMARY:
FemmeJock is a pelvic floor support system developed by pelvic floor physiotherapists for patients with pelvic organ prolapse in order to ameliorate symptoms of pelvic floor pressure and discomfort. The device is a girdle to be worn on the outside of underwear. The device is machine washable and there are no documented risks with wearing it. This product is currently being used by pelvic floor physiotherapists and has been subjectively reported by individual accounts as being successful in improving pelvic floor symptoms. The efficacy of this product has not been previously studied in women with pelvic organ prolapse. The investigators are proposing a pilot study with the following specific aims:

1. to assess patient satisfaction and continuation of use of the FemmeJock support system after 3 months of treatment.
2. to describe, if any, the reasons for discontinuation associated with the use of this product, and
3. to assess whether women experience improvement of pelvic floor symptoms after using this product.

DETAILED DESCRIPTION:
This will be a prospective pilot study in order to determine the efficacy and tolerability of FemmeJock in patients with pelvic organ prolapse. We plan to enroll 30 patients who will be recruited from the OU Health Science Center. We will offer study participation to patients who meet the inclusion criteria listed below, and who are: (1) awaiting surgical management and desire a temporary nonsurgical option, (2) seeking permanent nonsurgical treatment, or (3) who have a contraindication to surgical management.

ELIGIBILITY:
Inclusion Criteria:

* Pelvic organ prolapse, > stage II
* 1 or more prolapse associated symptoms:

  * Herniation symptoms
  * Pelvic pressure
  * Bulging tissue
  * Sexual dysfunction
* Patient willingness to enroll
* Available for 3 months of follow-up

Exclusion Criteria:

* Pregnancy or planning pregnancy within the next 3 months
* Perineal ulcers or trauma
* Anticipating relocation in next 3 months
* Current pessary use
* Dementia or inability to complete questionnaires
* Chronic inflammatory or infectious vulvar condition (i.e., dermatologic conditions: lichen sclerosis or lichen planus, or vulvar candidiasis)

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
to assess patient satisfaction and continuation of use of the FemmeJock support system after 3 months of treatment. | 2 years

SECONDARY OUTCOMES:
To describe, if any, the reasons for discontinuation associated with the use of this product. | 2 years
To assess whether women experience improvement of pelvic floor symptoms after using this product. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Lieschen H. Quiroz, M.D., Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States